CLINICAL TRIAL: NCT00859508
Title: A Prospective, Multi-Center, Randomized, Controlled Clinical Study Comparing SyntheCelTM Dura Replacement to Other Dura Replacements in Patients Requiring Dura Repair Following Cranial Surgery
Brief Title: Study of SyntheCelTM Dura Replacement to Other Dura Replacements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SyntheCel; NCT00454844 (obsolete NCT alias)
Record Dates: First submitted 2009-03-06; First posted 2009-03-11 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Cranial Dura Repair
Keywords: dura repair following cranial surgery

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- SyntheCel (Experimental)
  Interventions: Device: SyntheCel
- other FDA cleared dura replacements (Active Comparator)
  Interventions: Device: Other FDA cleared dura replacements

INTERVENTIONS:
Device: SyntheCel — Patients will be clinically followed post-surgery until hospital discharge or within ten (10) days of the procedure and at one (1) month, three (3) months and six (6) months. The data up to and including the 6 month follow-up visit will be used in demonstrating the performance of SyntheCelTM Dura Replacement.
  Arms: SyntheCel
Device: Other FDA cleared dura replacements — Patients will be clinically followed post-surgery until hospital discharge or within ten (10) days of the procedure and at one (1) month, three (3) months and six (6) months. The data up to and including the 6 month follow-up visit will be used in demonstrating the performance of SyntheCelTM Dura Replacement.
  Other Names: Duraform Dural Graft Implant; Duragen II Dural Regeneration Matrix; Duragen Dural Graft Matrix; Durepair Dura regeneration Matrix
  Arms: other FDA cleared dura replacements

SUMMARY:
Primary Objective: To demonstrate that the SyntheCelTM Dura Replacement performs similarly to or is substantially equivalent to other dura replacements for the repair of the cranial dura in patients undergoing surgical repair of the cranial dura.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 75 years of age
* Patient is scheduled for an elective cranial procedure requiring a dural incision
* Patient has an MRI no earlier than two months prior to the date of enrollment
* Surgical wound is expected to be Class I/clean
* Patient is available and willing to participate in the investigation for the duration of the study
* Patient has signed a written Informed Consent to participate in the study prior to any study mandated determinations or procedures. This does not include MRIs that may be performed prior to obtaining informed consent.

Exclusion Criteria:

* Patient has a cranial metallic implant(s) that would interfere with evaluation of the device or recovery
* Patient is somnolent or comatose (Glasgow score< 8)
* Patient has had a prior intracranial neurosurgical procedure in the same anatomical location
* Patient will require use of a dural adhesive or sealant
* Patient has known hydrocephalus
* Patient's life expectancy is less than 6 months
* Patient has a systemic infection (e.g. urinary tract infection (UTI), active pneumonia) or evidence of any surgical site infection, fever > 101°F, positive blood culture and/or a positive chest x-ray for acute infectious process
* Patient has known allergy to device component (cellulose)
* Patient is an acute cranial trauma surgical case
* Patient has a local cranial infection
* Patient has had chemotherapy and/or radiation treatment within 12 weeks prior to surgery, or has chemotherapy and/or radiation treatment planned 10 weeks post surgery
* Patient has been clinically diagnosed with malignancy (other than basal cell carcinoma or low grade glioma), uncontrolled diabetes, sepsis, systemic collagen disease
* Patient has creatinine levels > 2.0 mg/dL
* Patient has total bilirubin level > 2.5 mg/dL
* Patent has clinically significant coagulopathy with a partial thromboplastin time (PTT) ≥ 35, international normalized ratio (INR) ≥ 1.2, or is receiving Warfarin or Coumadin
* Patient has a compromised immune system or autoimmune disease (white blood cell (WBC) count <4000/uL or >20,000/uL)
* Patient is participating in another clinical trial using investigational devices/drugs
* Patient is pregnant or breastfeeding or wishes to become pregnant during the course of the study
* Patient is unable or unwilling to sign a consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Barrow Neurosurgical Institute, Scottsdale, Arizona
  - Stanford Medical Center, Stanford, California
  - University of Florida, Gainesville, Florida
  - Oregon Health Sciences University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Texas, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University School of Medicine, Morgantown, West Virginia

REFERENCES:
- [Result] Rosen CL, Steinberg GK, DeMonte F, Delashaw JB Jr, Lewis SB, Shaffrey ME, Aziz K, Hantel J, Marciano FF. Results of the prospective, randomized, multicenter clinical trial evaluating a biosynthesized cellulose graft for repair of dural defects. Neurosurgery. 2011 Nov;69(5):1093-103; discussion 1103-4. doi: 10.1227/NEU.0b013e3182284aca. PMID 21670715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was approved to enroll subjects from a maximum of 10 US medical institutions (public and academic research center hospitals). Subjects were enrolled from February 2006 to June 2008.
Pre-assignment Details: A total of 105 patients that initially met the inclusion/exclusion criteria were enrolled and randomized. Of those 105 patients, 99 received surgical treatment. Of those not treated, reasons included: change in diagnosis, not meeting Inclusion/Exclusion criteria, subject voluntary withdrawl, and investigator decision.
Groups:
- SyntheCel: The investigational group consists of patients who received the SyntheCel Dura Replacement device.
- Other FDA Cleared Dura Replacements: The Control group consists of other dura replacements that have been cleared for marketing by the FDA, including: Duraform Dural Graft Implant, Duragen II Dural Regeneration Matrix, Duragen Dural Graft Matrix, and Durepair Dura regeneration Matrix.
Period: Overall Study
Arm/Group | SyntheCel | Other FDA Cleared Dura Replacements
Started | 68 | 37
Completed | 62 | 37
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SyntheCel | Other FDA Cleared Dura Replacements | Total
Number analyzed (Participants) | 68 | 37 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 31 | 92
  >=65 years | 7 | 6 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.85) | 48.6 (14.03) | 47.2 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 25 | 75
  Male | 18 | 12 | 30
Region of Enrollment [Number; unit: participants]
  United States | 68 | 37 | 105

OUTCOME MEASURES:

1. Primary Outcome: Absence of Cerebrospinal Fluid (CSF) Fistula and Pseudomeningocele
Description: The primary endpoint for measuring effectiveness is such that an individual patient's treatment success requires the absence of CSF fistula (drainage from wound or sinus) and pseudomeningocele within 6 months post-operatively confirmed by radiographic evaluation and physical examination of the surgical site.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | SyntheCel | Other FDA Cleared Dura Replacements
Number analyzed (Participants) | 59 | 34
participants | 57 | 33

2. Secondary Outcome: Modified Rankin Scale (Patient Function Assessment)
Time Frame: up to 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Assessment of Changes in Body Systems (e.g., Head, Neurovascular, Etc.)
Time Frame: up to 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Wound Healing Assessment
Time Frame: up to 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Device Handling Characteristics (i.e., Ease of Use, Strength, Suturability, Seal Quality)
Time Frame: up to 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Radiographic Evaluation
Description: Radiographic evaluation (to determine the presence or absence of the following at the 6 month follow-up visit)
  * Adhesion formation
  * Membrane formation
  * Abnormal thickening along graft (device implant) site
  * Brain edema adjacent to graft (device implant) site
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SyntheCel | Other FDA Cleared Dura Replacements
Serious Adverse Events (participants affected / at risk) | 23/62 | 9/37
Other Adverse Events (participants affected / at risk) | 57/62 | 30/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyntheCel (N=62) | Other FDA Cleared Dura Replacements (N=37)
ANEMIA (Blood and lymphatic system disorders) | 2 | 0
BRAIN EDEMA (Nervous system disorders) | 2 | 0
CARDIOVASCULAR (Cardiac disorders) | 0 | 1
CSF LEAK (Nervous system disorders) | 2 | 0
DEATH (General disorders) | 0 | 1
DRUG REACTION (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL (Gastrointestinal disorders) | 2 | 0
HEADACHE (General disorders) | 2 | 0
HEMORRHAGE (Vascular disorders) | 1 | 0
HYDROCEPHALUS (Nervous system disorders) | 2 | 1
INFECTION-OTHER (Infections and infestations) | 1 | 0
INFECTION-SURGICAL SITE DEEP (Infections and infestations) | 1 | 0
INFECTION-SURGICAL SITE SUPERFICIAL (Infections and infestations) | 1 | 1
MUSCULOSKELETAL (Musculoskeletal and connective tissue disorders) | 1 | 0
NEUROLOGICAL (Nervous system disorders) | 7 | 1
PAIN (General disorders) | 1 | 0
PARESTHESIA (Nervous system disorders) | 1 | 1
PSYCHOLOGICAL (Psychiatric disorders) | 1 | 0
RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 2 | 2
STROKE (Vascular disorders) | 2 | 1
SURGERY-OTHER (Surgical and medical procedures) | 2 | 2
SURGERY-REOPERATION (INDEX SITE) (Surgical and medical procedures) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyntheCel (N=62) | Other FDA Cleared Dura Replacements (N=37)
ANEMIA (Blood and lymphatic system disorders) | 1 | 1
BRAIN EDEMA (Nervous system disorders) | 0 | 1
CARDIOVASCULAR (Cardiac disorders) | 5 | 7
CSF LEAK (Nervous system disorders) | 1 | 0
DEATH (General disorders) | 0 | 0
DERMATOLOGICAL (Skin and subcutaneous tissue disorders) | 7 | 1
DIPLOPIA (Eye disorders) | 1 | 2
DIZZINESS (General disorders) | 10 | 2
DRUG REACTION (Injury, poisoning and procedural complications) | 9 | 6
EDEMA (General disorders) | 13 | 3
FATIGUE (General disorders) | 9 | 2
FEVER (Infections and infestations) | 4 | 1
GASTROINTESTINAL (Gastrointestinal disorders) | 18 | 11
GENITOURINARY (Renal and urinary disorders) | 1 | 0
HEADACHE (General disorders) | 25 | 11
HEMATOMA (Vascular disorders) | 1 | 1
HEMORRHAGE (Vascular disorders) | 0 | 0
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HYDROCEPHALUS (Nervous system disorders) | 0 | 0
INFECTION-OTHER (Infections and infestations) | 3 | 3
INFECTION-SURGICAL SITE DEEP (Infections and infestations) | 0 | 0
INFECTION-SURGICAL SITE SUPERFICIAL (Infections and infestations) | 2 | 1
INSOMNIA (General disorders) | 4 | 2
MUSCULOSKELETAL (Musculoskeletal and connective tissue disorders) | 8 | 4
NEUROLOGICAL (Nervous system disorders) | 27 | 14
OTHER (General disorders) | 16 | 5
PAIN (General disorders) | 12 | 13
PAIN-INCISION (Skin and subcutaneous tissue disorders) | 7 | 5
PARATHESIA (Nervous system disorders) | 4 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 1
PSYCHOLOGICAL (Psychiatric disorders) | 5 | 5
RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 3 | 4
SEIZURE (Nervous system disorders) | 3 | 0
SEROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0
STROKE (Vascular disorders) | 0 | 0
SUBDURAL HEMATOMA (Vascular disorders) | 1 | 1
SURGERY-REOPERATION (INDEX SITE) (Surgical and medical procedures) | 0 | 0
THROMBOSIS (Vascular disorders) | 1 | 0
URINARY TRACT INFECTION (Renal and urinary disorders) | 2 | 0
WOUND ISSUES-OTHER (Skin and subcutaneous tissue disorders) | 6 | 4
SURGERY-OTHER (Surgical and medical procedures) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less